CLINICAL TRIAL: NCT04986124
Title: A Survey of Quality of Life in Chinese Working and School Age Population With Major Depressive Disorder
Brief Title: Quality of Life in Chinese Working and School Age Population With MDD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Beijing HuiLongGuan Hospital (Other); Huaxi Hospital (Other); Second Xiangya Hospital of Central South University (Other); Nanjing Brain Hospital, Nanjing Medical University (Unknown); Guangzhou Psychiatric Hospital (Other Government); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-76
Record Dates: First submitted 2021-04-08; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder; Remission
Keywords: cognitive function; social function; quality of life; working and school age population
MeSH Terms: conditions — Depressive Disorder, Major; Social Adjustment | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDD patients: No intervention.
  Interventions: Other: treatment as usual

INTERVENTIONS:
Other: treatment as usual — No inervention. Treatment regime remains unchanged.

SUMMARY:
Major depressive disorder (MDD) is a common mental illness with high prevalence and global burden. Previous studies revealed that over 70% patients in remission still had decreased quality of life, severe function impairment, low positive mental health score and poor coping ability. However, few studies focus on working and school age patients with MDD. A GBD survey showed that over 40% MDD patients are 15-50 years old. Therefore, we initiate the present multi-center cross-sectional survey to investigate the associations between clinical symptoms, cognitive function, occupational/study ability, and quality of life in Chinese working and school age population with MDD who are in remission.

DETAILED DESCRIPTION:
This is a multi-center cross-sectional study. Patients with MDD who received medication treatment and achieved remission for at least 8 weeks will be enrolled. For all the participants, demographic information will be collected; clinical symptoms, cognitive function, occupational/study ability, and quality of life will be evaluated by using 17-items HAMD, PHQ-9, HAMA, PSQI, SHAPS, HCL-32, SDS, LEAPS, QOL-6, PFQ and THINC-it toolkit.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients;
* Men or women aged between 16 and 50, with junior high school education or above;
* According to medical history, patients should be diagnosed with major depressive episode by two or above psychiatric doctors based on ICD-10 criteria;
* According to assessment, patients should meet the DSM-5 criteria for MDD when in past episodes;
* Patients received stable ant-depression medication treatment for at least 8 weeks before enrolment;
* 17-item HAMD total score ≤ 7;
* Willing to participate in this study, and sign an informed consent.

Exclusion Criteria:

* HCL-32 total score < 12;
* Diagnosed with bipolar disorder;
* Suffering from some serious physical diseases (e.g. moderate or severe brain injury, central nervous system diseases, or other unstable physical condition affecting the whole body) adversely affects the performance on neuropsychological test or rating scales;
* Received ECT in the past 6 months.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with MDD in working and school age who recieved medication treatment and achieved remission for at leat 8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
The Sheehan disability scale (SDS) | up to 1 weeks
  To evaluate the functional impairment, including work/study, daily life and family responsibility. The score of each subscale ranged from 0 to 10 which means from no impairment to loss of function.
Quality of Life, short form 6 (QOL-6) | up to 4 weeks
  To evaluate the quality of life in patients with MDD. The higher the total score, the better the quality of life.
The Psychosocial Function Questionnaire in Patients with Depression (PFQ) | up to 1 weeks
  To evaluate the psychosocial function of patients with MDD. The lower total score means the severer psychosocial function impairment.

SECONDARY OUTCOMES:
The Lam Employment Absence and Productivity Scale (LEAPS) | up to 2 weeks
  To evaluate the work capacity. The higher total score means the severer impairment of work capacity.
The Hamilton Depression Scale-17 items (HAMD) | up to 1 weeks
  To evaluate the severity of depressive symptoms by clinicians. Remission: total score < 7.
Patient Health Questionnaire-9 (PHQ-9) | up to 2 weeks
  to evaluate the severity of depressive symptoms by patients. Remission: total score < 4.
The Hamilton Anxiety Scale (HAMA) | up to 1 weeks
  To evaluate the severity of anxiety symptoms by clinicians. The total score < 6: no anxiety sympotom.
Pittsburgh Sleep Quality Index (PSQI) | up to 4 weeks
  To evaluate the sleep quality. The lower the total score, the better sleep quality (<5).
The Snaith-Hamilton Pleasure Scale (SHAPS) | up to 4 weeks
  To evaluate the severity of anhedonia. The higher total score means the severer of anhedonia.
THINC-it toolkit | up to 1 weeks
  To assess the cognitive function in patients with MDD specifically. The composite THINC-it tool score is the integrated total score of results from performance on five sub-component cognitive tests of the THINC-it tool.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D., Ph.D, Principal Investigator — Shanghai Mental Health Center (SMHC)
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No